CLINICAL TRIAL: NCT07226843
Title: NOVA-BCL6-1, A First-in-Human, Multicenter Phase 1a/1b Study to Investigate Safety, Tolerability, Pharmacokinetics, and Efficacy of LY4584180 in Adult Participants With Previously Treated Hematologic Malignancies
Brief Title: A Study of LY4584180 in Adult Participants With Previously Treated Blood Cancers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27804; J6Y-OX-JBFA (Other: Eli Lilly and Company); 2025-523601-16-00 (Other: EU CTIS Number)
Record Dates: First submitted 2025-11-07; First posted 2025-11-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Lymphoma, Non-Hodgkin's; Lymphoma, Diffuse Large B-Cell; Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1a-Monotherapy Dose Escalation (Cohort A1) (Experimental): LY4584180 monotherapy administered orally
  Interventions: Drug: LY4584180
- Phase 1a-Optional Monotherapy Dose Optimization (Cohort A2) (Experimental): LY4584180 monotherapy administered orally
  Interventions: Drug: LY4584180
- Phase 1b-Dose Expansion-Monotherapy (Cohort B1-B4) (Experimental): LY4584180 monotherapy administered orally
  Interventions: Drug: LY4584180
- Phase 1b-Dose Expansion-Combination (Cohort B5) (Experimental): LY4584180 administered orally in combination with rituximab administered through IV infusion
  Interventions: Drug: LY4584180; Drug: Rituximab

INTERVENTIONS:
Drug: LY4584180 — administered orally
Drug: Rituximab — administered through IV infusion
  Arms: Phase 1b-Dose Expansion-Combination (Cohort B5)

SUMMARY:
The main purpose of this study is to evaluate safety and efficacy, and measure how much LY4584180 gets into the bloodstream and how long it takes the body to eliminate it in patients with previously treated blood cancers. For each participant, the study could last about 9 months or possibly longer including screening.

ELIGIBILITY:
Inclusion Criteria:

* Has been treated for the following blood cancers and has received at least 2 prior lines of systemic therapy or not eligible for available therapy:

  * Diffuse large B-cell lymphoma - not otherwise specified
  * High-grade B-cell lymphoma
  * Follicular large B-cell lymphoma
  * Follicular lymphoma
  * Other non-Hodgkin lymphoma
* Has measurable disease
* Has discontinued all previous treatments for cancer and has recovered from the immediate effects of therapy

Exclusion Criteria:

* Has an active second cancer
* Has known or suspected history of central nervous system involvement
* Has known Cytomegalovirus infection. Participants with negative status are eligible
* Has known hepatitis B or C infection or HIV
* Has significant heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Number of Dose-Limiting Toxicities (DLTs) and DLT-Equivalent Toxicities | Baseline up to Day 28
  Number of Dose-Limiting Toxicities (DLTs) and DLT-Equivalent Toxicities
Number of Participants with One or More Serious Adverse Events (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to 3 Years
  Number of Participants with One or More Serious Adverse Events (SAEs) Considered by the Investigator to be Related to Study Drug Administration
To Evaluate the Preliminary Antitumor Activity of LY4584180: Objective Response Rate (ORR) | Baseline up to 3 Years
  To Evaluate the Preliminary Antitumor Activity of LY4584180: Objective Response Rate (ORR)

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Serum Concentration (Cmax) of LY4584180 | Baseline to Day 8
  PK: Cmax of LY4584180
PK: Area Under the Concentration (AUC) Versus Time Curve of LY4584180 | Baseline to Day 8
  PK: AUC versus time curve of LY4584180

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (32):
- United States (19):
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - City of Hope, Duarte, California
  - University of California, Los Angeles (UCLA) - Medical Center, Los Angeles, California
  - University of California, San Francisco (UCSF) - Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Miami - Sylvester Cancer Center, Miami, Florida
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - University of Rochester, Rochester, New York
  - The Ohio State University (OSU), Columbus, Ohio
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology - DFW (Sammons CC), Dallas, Texas
  - University of Washington - Fred Hutchinson Cancer Center (Seattle Cancer Care Alliance), Seattle, Washington
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- France (2):
  - CHU de Nantes - Hotel-Dieu, Nantes
  - Institut Curie, Paris
- Germany (2):
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Frankfurt - Klinikum der Johann Wolfgang Goethe Universitaet, Frankfurt am Main
- Italy (2):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna - Policlinico di Sant Orsola, Bologna
  - Istituto Europeo di Oncologia, Milan
- Instytut Hematologii i Transfuzjologii w Warszawie, Warsaw, Poland
- Spain (2):
  - Institut Catala d'Oncologia - L'Hospitalet, Barcelona
  - South Texas Accelerated Research Therapeutics (START) Madrid - Hospital Fundacion Jimenez Diaz, Madrid
- United Kingdom (4):
  - King's College Hospital, London
  - Nottingham City Hospital, Nottingham
  - Derriford Hospital, Plymouth
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No